CLINICAL TRIAL: NCT03550586
Title: Long Term Outcomes of Parturients Suffering From a Post Dural Puncture Headache Following an Accidental Dural Puncture (PDPH)
Brief Title: Long Term Outcomes Following a Post Dural Puncture Headache
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0536-17-RMC
Record Dates: First submitted 2018-04-22; First posted 2018-06-08 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2018-04

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parturients suffering from a PDPH: Parturients suffering form a PDPH following an accidental dural puncture between the years 2007-2017 will be contacted by phone and verbal consent will be obtained for participation in the study. All participants will be requested to answer an IRB approved telephone script. Parturients will be assed for postpartum depression using the Edinburgh Postnatal Depression Scale (EPDS) translated into Hebrew . They will also be assed for PTSD using the validated PTSD questionnaire.Additionally in order to examine long term risk for chronic pain and backache parturients will be assed for persistent pain using the validated Brief Pain Inventory questionnaire ,and the validated Oswestry low back pain questionnaire
  Interventions: Other: Questionaires
- Parturients not suffering from a PDPH: This group will consistent of a control group of women receiving epidural analgesia on the same day as those women who suffered an ADP. This participants will be contacted by phone and verbal consent will be obtained for participation in the study. All participants will be requested to answer an IRB approved telephone script. Parturients will be assed for postpartum depression using the Edinburgh Postnatal Depression Scale (EPDS) translated into Hebrew . They will also be assed for PTSD using the validated PTSD questionnaire.Additionally in order to examine long term risk for chronic pain and backache parturients will be assed for persistent pain using the validated Brief Pain Inventory questionnaire ,and the validated Oswestry low back pain questionnaire
  Interventions: Other: Questionaires

INTERVENTIONS:
Other: Questionaires — Parturients will be assed for postpartum depression using the Edinburgh Postnatal Depression Scale (EPDS)translated into Hebrew . They will also be assed for PTSD using the validated PTSD questionnaire . Additionally in order to examine long term risk for chronic pain and backache parturients will be assed for persistent pain using the validated Brief Pain Inventory questionnaire ,and the validated Oswestry low back pain questionnaire .

SUMMARY:
Epidural analgesia is considered a gold standard method for treatment of labor pain. One of the major risks with epidural analgesia is an accidental dural puncture, which leads to a post dural puncture headache. This headache is associated with significant maternal morbidity and can result in severe maternal consequences.

Post traumatic stress disorder (PTSD) is defined as an anxiety syndrome, resulting from a traumatic experience. Postpartum PTSD, is a form of PTSD that can occur in relation to a traumatic birth experience. As PDPH is unexpected and can cause severe maternal sequele, PDPH can exhibit a posttraumatic stress response. Therefore we hypothesize that parturients who suffered from a PDPH are at higher risk for developing PP-PTSD.

To date, very few reports have examined the long term outcomes of parturients suffering from a PDPH. As a follow up to the national survey of PDPH management in Israel the investigators aim, in this prospective multi center, observational study, to evaluate the long term outcomes of parturients suffering from a PDPH, including chronic headache, backache, postpartum depression, decreased breastfeeding and the development of PP PTSD.

DETAILED DESCRIPTION:
Introduction:

Epidural analgesia is considered a gold standard method for treatment of labor pain . However one of the major risks with epidural analgesia is an accidental dural puncture, a common complication occurring in 0.4-6% of the obstetric population . ADP increases the risk of developing a post dural puncture headache (PDPH) in 50% of parturients. PDPH is defined as a postural headache that worsens within fifteen minutes of standing and is relieved in the supine position . PDPH results from a CSF leakage from the intrathecal space, causing a decrease in CSF volume and pressure .

PDPH is associated with significant maternal morbidity, prolonging hospital stay, preventing ambulation and impairing maternal neonatal bonding . Less frequently PDPH can cause severe maternal complications resulting in posterior reversible encephalopathic syndrome , pneumocephalus , or a subdural hematoma .

Treatment protocols for PDPH vary greatly, with numerous existing conservative/ invasive treatment options . Conservative treatment includes bed rest, fluids administration, non-steroidal anti-inflammatory drugs and caffeine intake. The most standard invasive method for treatment of PDPH with a reported success rate of 70-90% includes the epidural blood patch (EPD) which is applied by injecting autologous blood epidurally .

Several factors have been found to increase the risk for developing a PDPH and increasing the duration of a PDPH including young age, low BMI and previous history of anxiety or depression .

Posttraumatic stress disorder is classified as an anxiety syndrome one may develop in response to a traumatic experience. Clinical manifestations include persistent re-experience, avoidance of traumatic memories, hyperarousal and emotional numbing . In a retrospective analysis war related PTSD was not associated with increased risk of PDPH.

Post partum (PP) PTSD is a form of PTSD occurring in the postpartum period in relation to a traumatic birth . As PDPH is unexpected and can cause severe maternal sequele, PDPH can exhibit a posttraumatic stress response. Therefore the investigators hypothesize that parturients who suffered from a PDPH are at higher risk for developing PP-PTSD.

To date very few reports have examined the long term outcomes of parturients suffering from a PDPH associated with epidural analgesia. In a prospective, case control trial Webb et al demonstrated an increased risk for developing a chronic headache and backache in 40 parturients who suffered an accidental dural puncture with a large gauge needle . In a five year follow-up study examining long term consequences of PDPH, PDPH was associated with persistent headache and backache in the obstetric population. In a case control trial evaluating long term auditory function following EBP treatment for PDPH, a minor hearing loss was detected in the PDPH group . However, these studies had a small sample size.

As a follow up to the national survey of PDPH management in Israel the investigators aimed in this study to evaluate the long term consequences of PDPH including chronic headache, backache, postpartum depression (PPD), decreased breastfeeding and the development of PP PTSD.

Study Objective:

In this study the investigators intend to evaluate the long term sequelae of parturients who suffered from an accidental dural puncture and a subsequent PDPH.

Primary Aims:

This study's primary objective is to examine whether parturients suffering from a PDPH are at higher risk long-term for developing PP-PTSD than their counterparts.

Secondary aims:

Secondary aims include long term outcomes of parturients who suffered from PDPH:

* Chronic headache
* Chronic backache
* Comparing long term outcomes of parturients suffering from a PDPH with conservative treatment verses epidural blood patch treatment.
* PPD
* Breastfeeding outcomes including duration of breastfeeding
* Women will also be questioned about other labor experiences including analgesic consumption, breastfeeding outcome.

Study Design This study is a prospective multi center cohort, study. Following obtaining approval from the local Institutional Review Board at each center, all women who developed a PDPH following an ADP between the years 2007-2017 will be contacted by phone and verbal consent will be obtained for participation in the study. Each participant will be compared to two women receiving epidural analgesia on the same day as those women who suffered an ADP. All participants will be requested to answer an IRB approved telephone script. Parturients will be assed for postpartum depression using the Edinburgh Postnatal Depression Scale (EPDS)translated into Hebrew . They will also be assed for PTSD using the validated PTSD questionnaire . Additionally in order to examine long term risk for chronic pain and backache parturients will be assed for persistent pain using the validated Brief Pain Inventory questionnaire ,and the validated Oswestry low back pain questionnaire . Parturients will also be asked about other labor experiences including analgesic consumption and breastfeeding outcome, in cases of breastfeeding cessation women will be asked an open-ended question about the reason for discontinuation.

Data collection:

Additional data will be collected from an electronic medical file database. Data collection will include; parturient's demographic data, obstetric data, in case of EBP treatment procedural data (level of injection, volume of blood injected, loss of resistance technique- air/saline, anesthesiologist experience, time of procedure, duration of procedure, technical difficulties, visual analogue score (VAS) upon lying down/ upon sitting up - before the EBP and upon release

ELIGIBILITY:
Inclusion Criteria:

- All cases of parturients suffering from a PDPH during the years 2007-2017.

Exclusion Criteria:

- Women unable to be answer a questionnaire in Hebrew. Women under the age 18 Women suffering from a PDPH following spinal anesthesia for cesarean section.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All women who developed a PDPH following an ADP between the years 2007-2017 at rabin medical center and at Assaf Harofeh Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder (PTSD) questionnaire score | Up to ten years postpartum (Answer at telephone survey)
  The total PTSD questionnaire score using the validated PTSD questionnaire

SECONDARY OUTCOMES:
The total Edinburgh Postnatal Depression Scale (EPDS) questionnaire score | Up to ten years postpartum (Answer at telephone survey)
  Parturients will be assed for postpartum depression using the Edinburgh Postnatal Depression Scale
The total score on the Brief Pain Inventory questionnaire | Up to ten years postpartum (Answer at telephone survey)
  Parturients will be assed for chronic pain using the validated Brief Pain Inventory questionnaire questionnaire
The total score on the Oswestry low back pain questionnaire | Up to ten years postpartum (Answer at telephone survey)
  Parturients will be assed for back pain using the validated Oswestry low back pain questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sharon O Zinger, Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Dr. Chatuib Zoya, Be’er Ya‘aqov
  - Beilinson hospital, Petach Tikvah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradbury CL, Singh SI, Badder SR, Wakely LJ, Jones PM. Prevention of post-dural puncture headache in parturients: a systematic review and meta-analysis. Acta Anaesthesiol Scand. 2013 Apr;57(4):417-30. doi: 10.1111/aas.12047. Epub 2012 Dec 28. PMID 23278515
- [Background] Sachs A, Smiley R. Post-dural puncture headache: the worst common complication in obstetric anesthesia. Semin Perinatol. 2014 Oct;38(6):386-94. doi: 10.1053/j.semperi.2014.07.007. Epub 2014 Aug 19. PMID 25146108
- [Background] Arevalo-Rodriguez I, Ciapponi A, Roque i Figuls M, Munoz L, Bonfill Cosp X. Posture and fluids for preventing post-dural puncture headache. Cochrane Database Syst Rev. 2016 Mar 7;3(3):CD009199. doi: 10.1002/14651858.CD009199.pub3. PMID 26950232
- [Background] Angle P, Tang SL, Thompson D, Szalai JP. Expectant management of postdural puncture headache increases hospital length of stay and emergency room visits. Can J Anaesth. 2005 Apr;52(4):397-402. doi: 10.1007/BF03016283. PMID 15814755
- [Background] Webb CA, Weyker PD, Zhang L, Stanley S, Coyle DT, Tang T, Smiley RM, Flood P. Unintentional dural puncture with a Tuohy needle increases risk of chronic headache. Anesth Analg. 2012 Jul;115(1):124-32. doi: 10.1213/ANE.0b013e3182501c06. Epub 2012 Mar 30. PMID 22467897
- [Background] Shah R, Kubisz-Pudelko A, Reid J. Posterior reversible encephalopathy syndrome following an inadvertent dural puncture during an emergency laparotomy for ischemic colitis - a case report. Local Reg Anesth. 2014 Jan 20;7:1-4. doi: 10.2147/LRA.S57660. eCollection 2014. PMID 24600245
- [Background] Gomez-Rios MA, Fernandez-Goti MC. Pneumocephalus after inadvertent dural puncture during epidural anesthesia. Anesthesiology. 2013 Feb;118(2):444. doi: 10.1097/ALN.0b013e31825e6ecc. No abstract available. PMID 22692380
- [Background] Liang MY, Pagel PS. Bilateral interhemispheric subdural hematoma after inadvertent lumbar puncture in a parturient. Can J Anaesth. 2012 Apr;59(4):389-93. doi: 10.1007/s12630-011-9664-6. Epub 2012 Jan 4. PMID 22215524
- [Background] Basurto Ona X, Uriona Tuma SM, Martinez Garcia L, Sola I, Bonfill Cosp X. Drug therapy for preventing post-dural puncture headache. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD001792. doi: 10.1002/14651858.CD001792.pub3. PMID 23450533
- [Background] Stannard D. Epidural blood patching for preventing and treating postdural puncture headache. J Perianesth Nurs. 2011 Dec;26(6):411-2. doi: 10.1016/j.jopan.2011.09.002. No abstract available. PMID 22099135
- [Derived] Orbach-Zinger S, Eidelman LA, Livne MY, Matkovski O, Mangoubi E, Borovich A, Wazwaz SA, Ioscovich A, Zekry ZHB, Ariche K, Weiniger CF. Long-term psychological and physical outcomes of women after postdural puncture headache: A retrospective, cohort study. Eur J Anaesthesiol. 2021 Feb 1;38(2):130-137. doi: 10.1097/EJA.0000000000001297. PMID 32858584